CLINICAL TRIAL: NCT00302809
Title: Effect of Concord Grape Juice on Blood Pressure and Vascular Function in Subjects With Pre-Hypertension and Stage 1 Hypertension
Brief Title: Blood Pressure Lowering Effects of Grape Juice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Welch's, Inc. (Industry)
Responsible Party: Joseph A. Vita, MD, Boston University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-24568
Record Dates: First submitted 2006-03-13; First posted 2006-03-15 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Hypertension
Keywords: Flavonoids; Arterial stiffness; Blood pressure; Endothelium; Inflammation
MeSH Terms: conditions — Hypertension; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Concord Grape Juice — Approximately 16 oz of grape juice or placebo

SUMMARY:
Recent studies suggest that a diet rich in fruit and vegetables can lower blood pressure, and a number of lines of evidence suggest that grape products may have such an effect. The purpose of this study is to determine whether consuming grape juice lowers blood pressure in individuals with pre-hypertension or stage I hypertension.

DETAILED DESCRIPTION:
Elevated blood pressure (BP) is among the most common and important risk factors for atherosclerosis. A number of non-pharmacological therapies have successfully been applied to prevent the development of elevated BP or reduce elevated BP. For example the DASH Study showed that a diet rich in fruits, vegetables and low fat dairy products, and reduced in saturated fat, total fat and cholesterol, substantially lowered blood pressure in normotensive and hypertensive individuals.

Within the past three years a number of small clinical trials have suggested suggest that drinking purple grape juice for a period of 6-12 weeks may lower blood pressure individuals with elevated blood pressure. Other clinical trials have shown that Concord grape juice improves the function of the vascular endothelium, possibly providing an explanation for the beneficial effect. However, there is a need for a prospective, controlled study to determine whether grape juice has a beneficial effect on blood pressure.

The present study will compare the effect of drinking Concord purple grape juice (7 ml/kg or about 16 oz/day for a 70 kg person) and the effect of calorie-matched placebo on 24-hour ambulatory blood pressure, blood pressure reactivity, and vascular function in men and women in the category of "pre-hypertension" (defined as blood pressure greater than 120/80, but less than 149/89 mmHg and Stage 1 hypertension (defined as blood pressure greater than 140/90, but less than 160/100). This study will specifically recruit patients with systolic blood pressure of 130-159 mmHg or diastolic blood pressure of 85-99 mmHg. The study will be double blind and have a crossover design with the order of treatment randomized (grape juice first or placebo first). A dietician will provide all subjects with formal instruction in a low salt diet, which is the current recommended initial therapy for patients with Stage 1 hypertension.

After a 1-week run-in period, subjects will consume each beverage for 8 weeks with a 4-week rest period between treatments. Blood pressure will be measured before and after each treatment period using a 24-hour ambulatory blood pressure recording. After each treatment period, we will measure changes in blood pressure induced by psychological challenge (mental arithmetic and computer tasks) and by the cold pressor test. In order to gain insight into the potential mechanisms of benefit, we will also examine the effects of beverage consumption on endothelial function, stiffness of the central aorta, fasting glucose and insulin, body weight, and markers of systemic inflammation, including CD40 ligand and C-reactive protein. Finally, we will store plasma samples for future investigation of other potential effects of grape juice on the cardiovascular system.

We hypothesize that Concord grape juice will have favorable effects on blood pressure compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females
2. Body Mass Index (BMI) of less than 35.0 kg/m2
3. Systolic blood pressure (130-159 mmHg) and/or diastolic blood pressure (85-99 mm Hg) on two screening visits
4. Subject must be judged to be in good health on the basis of medical history; 5. Subject must not be taking any antihypertensive medications for at least one month prior to the Screening Visit

Exclusion Criteria:

1. History of clinically defined coronary artery disease, peripheral artery disease, stroke, active gastrointestinal ulcers, renal, or hepatic disease;
2. History of bleeding disorders or malabsorption syndromes;
3. Taking drugs for regulating hemostasis, including stable-dose aspirin;
4. History of active cancer
5. Females who are pregnant or planning to become pregnant
6. Use of weight-loss drugs (including over-the-counter and dietary supplements)
7. Diagnosed diabetes mellitus
8. Subjects who consume a vegetarian diet
9. Recent history (within the past 6 months) of alcohol or substance abuse.
10. Laboratory values outside the following ranges: serum potassium (3.5-5.1 mg/dl), creatinine (0.5-1.3 mg/dl), hematocrit (36-50%), white blood count (4.0-11.0 K/ul), platelet count (150-400 k/ul)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-03; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Blood pressure measured by 24-hour recorder | 8 weeks

SECONDARY OUTCOMES:
Pulse wave velocity | 8 weeks
Pulse amplitude tonometry | 8 weeks
Blood pressure during mental tasks | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Vita, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Dohadwala MM, Hamburg NM, Holbrook M, Kim BH, Duess MA, Levit A, Titas M, Chung WB, Vincent FB, Caiano TL, Frame AA, Keaney JF Jr, Vita JA. Effects of Concord grape juice on ambulatory blood pressure in prehypertension and stage 1 hypertension. Am J Clin Nutr. 2010 Nov;92(5):1052-9. doi: 10.3945/ajcn.2010.29905. Epub 2010 Sep 15. PMID 20844075